CLINICAL TRIAL: NCT06310460
Title: Prospective Monocentric Cohort Study to Evluate Pre-cut Papillectomy in Patients With Difficult Biliary Cannulation During Endoscopic Retrograde Cholangiopancreaticography
Brief Title: Evaluation of "PreCut-Papillectomy" in Difficult Biliary Cannulation
Status: Not yet recruiting | Type: Observational
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: PCP
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Papillectomy — Papillectomy prior to bile duct cannulation during ERCP

SUMMARY:
To evaluate the effectiveness and sefety of papillectomy to enable bile duct access during endoscopic retrograde cholangiography in patients with difficult biliary cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Difficult cannulation of bile duct

Exclusion Criteria:

* post-surgical upper GI anatomy
* previous endoscopic retrograde cholangiopancreaticography or percutaneous transhepatic cholangiography
* papilla within a diverticulum
* coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ERCP with intented bile duct cannulation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment success | During endoscopy
  Rate of successful cannulation of the bile duct after PreCut-papillectomy
Adverse event rate | Up to 30 days
  Rate of adverse events, as classifed by ASGE classification

IPD SHARING:
Plan to Share IPD: No